CLINICAL TRIAL: NCT05922735
Title: Seroprevalence of Monkeypox Infection Among People Living With HIV and PrEP Users
Acronym: MonVIP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: INSERM UMR S 1136 (Other); Institut de Recherche en Santé Publique, France (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: ANRS 0297s MonVIP
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Monkey Pox; HIV Infections
Keywords: Mpox; PrEP; HIV Infections; Mpox serology; Sexual behaviors
MeSH Terms: conditions — Mpox, Monkeypox; HIV Infections; Coitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population living with HIV and PrEP users: Population of people living with HIV and PrEP users followed in the infectious disease departments in Ile de France and in the province.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Serology from remaining blood sample Self-questionnaire about sexual behavior during the epidemy mpox

SUMMARY:
This is a cohort, non-health product, non-interventional biomedical research, multi-centric, to determine the seroprevalence of mpox infection in the population of people living with HIV and in PrEP users in Ile-de-France and in the province.

DETAILED DESCRIPTION:
The target population is the population of people living with HIV (PLHIV) (n=18,500) and PrEP users (n=4930) followed up in Parisian infectious and tropical diseases departments (SMIT) of the Pitié-Salpêtrière, Tenon, Saint-Antoine, Bichat, Saint-Louis, Necker hospitals, the University Department of Infectious and Traveller Diseases of Hôpital Dron (Tourcoing), the 190 health center, and the Maison de santé du Chemin vert (Paris).

The principal objective is to determine the seroprevalence of Monkeypox infection in the population of PLHIV and PrEP users followed in the infectious and tropical disease departments in 9 centers.

In addition to the primary objective, there exist the following secondary objectives:

* To assess the level of anti-Mpox antibodies in PLHIV and PrEP users
* To assess the level of anti-Mpox antibodies in PLHIV and PrEP users with a previous confirmed diagnosis of Mpox or if they have been recently vaccinated
* Assess antibody levels in PLHIV in relation to CD4 cell count and HIV viral load
* Study antibody kinetics and persistence over time (D0 (between November 1, 2021 and April 30, 2022), M6, M12)
* Study the Mpox seroconversion rate over time
* Determine the neutralizing activity of anti-Mpox antibodies in individuals with positive anti-Mpox ELISA serology.
* Describe the natural history of the disease, the different forms of the disease, their clinical characterization
* Describe sexual behavior and the impact of this health crisis on different aspects of their lives using a self-administered questionnaire
* To determine the prevalence of asymptomatic infections
* Proportion of participants with positive Mpox serology without PCR confirmed diagnosis
* History of childhood or recent smallpox vaccination

During the patient's follow-up consultation, after information and in the absence of an expression of no objection, inclusion will consist of recovering a blood sample taken between November 2021 and April 2022 during the HIV infection assessment or PrEP follow-up (no additional sample) and possibly the blood sample taken at M6 and/or M12 if this follow-up consultation has already taken place.

An online self-questionnaire will also be proposed to the patient (male only). It will be constructed from questions already validated in other surveys (Rapport au Sexe, Prévenir, Parcours).

A check on the appearance or persistence of antibodies will be carried out at M6 +/- 8 weeks and/or M12 +/- 8 weeks on tube bottoms of samples always taken as part of the HIV infection assessment or PrEP follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* People Living with HIV or PrEP users with a blood test within 6 months before the start of the epidemic (i.e. between 1/11/2021 and 30/04/2022, D0) and with a blood test scheduled at M6 and/or at M12 of this collection depending on the care, in the centers participating in the study
* Having been informed about the study and not having expressed his opposition
* Affiliated to a social security system or entitled person, AME beneficiary

Exclusion Criteria:

* Refusal of participation by the patient
* Under legal protection (guardianship/guardianship)
* Not able to understand the information and/or express opposition and/or not speaking French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is the population of PLHIV (n=18,500) and PrEP users (n=4930) followed up in the infectious and tropical diseases departments (SMIT) in 9 centers in Ile de France and province.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Mpox serology | 12 months
  The primary endpoint will be to determine the presence or not of anti-Mpox antibodies in the population of PLHIV or PrEP users

SECONDARY OUTCOMES:
Anti-Mpox antibodies | 12 months
  To determine the presence or not of anti-Mpox antibodies by ELISA in PLWHIV and PrEP users with a previous confirmed diagnosis of Mpox or with a recent vaccination
Antibody level in PLWHIV | 12 months
  Comparison of Mpox serology with CD4 count and viral load of PLHIV
Antibody kinetics | 12 months
  Comparison of Mpox antibody levels between D0, M6 and M12
Mpox seroconversion | 12 months
  Comparison of anti-Mpox serology results between D0, M6 and M12
Neutralizing activity | 12 months
  Observation of the number of serum-neutralization test results for all Mpox-positive samples
Natural history of Mpox | 12 months
  Collect information on date of seropositivity, date of onset of symptoms, types of symptoms, clinical features of infection.
Asymptomatic infections | 12 months
  Comparison of the proportion of asymptomatic vs. symptomatic in HIV-positive patients.
Mpox serology and PCR | 12 months
  Comparison of the proportion of asymptomatic, the proportion with symptoms without PCR confirmation, proportion vaccinated in the past or recently
Childhood or recent smallpox vaccination | 12 months
  Comparison of proportion with PCR-confirmed Mpox, proportion previously or recently vaccinated.
Sexual behavior | 12 months
  To count and collection of sexual behavior and impact of health crisis among PLWHIV and PrEP users via self-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Valérie POURCHER, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No